CLINICAL TRIAL: NCT01383668
Title: Combined PKCiota and mTOR Inhibition for Treatment of Advanced Squamous Lung Cancer
Brief Title: Sirolimus and Gold Sodium Thiomalate in Treating Patients With Advanced Squamous Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: lack of access to study drug
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC102A; NCI-2011-00968 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-06-24; First posted 2011-06-28 (Estimated); Last update posted 2020-04-01 (Actual); Status verified 2012-12

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Squamous Cell Lung Cancer; Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Sirolimus; Gold Sodium Thiomalate; Polymerase Chain Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (enzyme inhibitor therapy) (Experimental): Patients receive sirolimus PO QD on days 1-28 and gold sodium thiomalate IM on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sirolimus; Drug: gold sodium thiomalate; Other: pharmacological study; Genetic: RNA analysis; Genetic: polymerase chain reaction

INTERVENTIONS:
Drug: sirolimus — Given PO
  Other Names: AY 22989; Rapamune; rapamycin; SLM
Drug: gold sodium thiomalate — Given IM
  Other Names: Aurolate; Myochrysine; sodium aurothiomalate
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Genetic: RNA analysis — Correlative studies
Genetic: polymerase chain reaction — Correlative studies
  Other Names: PCR

SUMMARY:
This phase I trial studies the side effects and best dose of sirolimus and gold sodium thiomalate when given together in treating patients with advanced squamous non-small cell lung cancer (NSCLC). Sirolimus and gold sodium thiomalate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To determine the maximally tolerated dose (MTD) of ATM (gold sodium thiomalate) plus sirolimus. SECONDARY OBJECTIVES: I. To describe the adverse event profile associated with this treatment combination. II. To preliminarily evaluate the response rate, time to progression, progression-free survival and overall survival of patients treated with this treatment combination. TERTIARY OBJECTIVES: I. To evaluate tumor biomarkers of protein kinase C (PKCι) and mammalian Target Of Rapamycin (mTOR) signaling activity as predictors of response to ATM/sirolimus therapy. II. To evaluate the use of surrogate biomarkers of PKCι and mTOR inhibition in peripheral blood lymphocytes (PBLs) to monitor response to ATM/sirolimus therapy. OUTLINE: This is a dose-escalation study. Patients receive sirolimus orally (PO) once daily (QD) on days 1-28 and gold sodium thiomalate intramuscularly (IM) on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Cohort I (Dose Escalation) only: must have histologic proof of an advanced, solid tumor that is now unresectable
* Cohort II (MTD) only
* Patients must have platinum-refractory NSCLC (platinum-refractory defined as either disease progression either during or within 6 months of completion of first-line platinum-based chemotherapy)
* Must have measurable disease
* Must have received at least one prior approved chemotherapeutic regimen unless there is no known, approved therapeutic regimen for their malignancy
* Must have evidence of disease progression within the preceding 6 months - Absolute neutrophil count (ANC) >= 1500/uL
* Platelets (PLT) >= 100,000/uL
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* (Serum glutamic oxaloacetic transaminase [SGOT]) aspartate aminotransferase (AST) / (serum glutamic pyruvic transaminase [SGPT]) alanine transaminase (ALT) =< 3 x ULN or (SGOT) AST / (SGPT) ALT =< 5 x ULN if liver involvement
* Creatinine =< 1.5 x ULN
* Fasting blood glucose =< 126 mg/dL
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0, 1 or 2
* Ability to provide informed consent
* Willingness to return to Mayo Clinic in Florida for follow-up
* Life expectancy >= 84 days (3 months)
* Willing to provide blood and tissue samples for correlative research purposes; Note: the goals of this study include assessment of the biologic effects of the agent being tested and are, therefore, contingent upon availability of the biologic specimens
* Women of childbearing potential only: negative (serum) pregnancy test done =< 7 days prior to registration

Exclusion Criteria:

* Known standard therapy for the patient's disease that is potentially curative or definitely capable of extending life expectancy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Any of the following prior therapies:
* Chemotherapy =< 28 days prior to registration
* Mitomycin C/nitrosoureas =< 42 days prior to registration
* Immunotherapy =< 28 days prior to registration
* Biologic therapy =< 28 days prior to registration
* Radiation therapy =< 28 days prior to registration
* Radiation to > 25% of bone marrow
* Bevacizumab =< 28 days prior to registration
* Failure to fully recover from acute, reversible effects of prior chemotherapy regardless of interval since last treatment
* New York Heart Association classification III or IV
* Known central nervous system (CNS) metastases or seizure disorder; patients with known brain metastases that have been successfully treated and stable for >= 6 months without requirement for corticosteroids and without seizure activity will be eligible
* Patients with known diabetes mellitus unless well-controlled (fasting blood sugar [FBS] =< 126mg/dL and hemoglobin [Hb]A1C =< 7.0)
* Receiving therapeutic anticoagulation with warfarin; NOTE: prophylactic anticoagulation (i.e., low dose warfarin) of venous or arterial access devices is allowed, provided that International Normalized Ratio (INR) < 1.5; therapeutic anti-coagulation with low molecular weight heparin is allowed at time of registration
* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown: - Pregnant women - Nursing women - Men or women of childbearing potential who are unwilling to employ adequate contraception - Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-Food and Drug Administration [FDA] approved indication and in the context of a research investigation)
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients (other than that related to the use of corticosteroids) including patients known to be human immunodeficiency virus (HIV) positive
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Cohort II Only: other active malignancy =< 5 years prior to registration; EXCEPTIONS: non-melanotic skin cancer or carcinoma-in-situ of the cervix; NOTE: If there is a history or prior malignancy, patient must not be receiving other cytotoxic or molecularly targeted therapeutics treatment for their cancer; patients receiving certain hormonal manipulations as part of their treatment may be allowed to continue at the discretion of the principal investigator (PI) (e.g. luteinizing hormone-releasing hormone [LHRH] analogs for prostate cancer); concurrent endocrine therapy for breast cancer will not be permitted
* History of myocardial infarction =< 168 days (6 months) or congestive heart failure requiring use of ongoing maintenance therapy for life threatening ventricular arrhythmias
* Known allergy to ATM (Aurothiomalate [gold sodium thiomalate]) or other gold compounds
* >= Grade 2 hypertriglyceridemia
* >= Grade 2 hypercholesterolemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2013-02-08 (Actual); Study Completion 2013-02-08 (Actual)

PRIMARY OUTCOMES:
Maximally tolerated dose (MTD) of ATM plus sirolimus | 28 days
  MTD is defined as the dose level below the lowest dose that induces dose-limiting toxicity (DLT) in at least one-third of patients (at least 2 of a maximum of 6 new patients). A total of 6 patients treated at the MTD will be sufficient to identify common toxicities at the MTD.

SECONDARY OUTCOMES:
To describe the adverse event profile associated with the treatment combination of ATM plus sirolimus. | Up to 3 months after completion of study treatment
Confirmed response rate | Every 6 weeks
Overall survival time | Up to 3 months after completion of study treatment
Progression-free survival (PFS) | Up to 3 months after completion of study treatment
Time-to-progression (TTP) | Up to 3 months after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael Menefee, Principal Investigator — Mayo Clinic